CLINICAL TRIAL: NCT05262101
Title: Single-arm, Open-label, Multicenter Phase Ib Clinical Trial of TQB2858 Injection in the Treatment of Advanced High-grade Sarcoma
Brief Title: Clinical Trial of TQB2858 Injection in the Treatment of Advanced High-grade Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor has decided to terminate this study based on the current clinical research status of dual antibody drugs and full communication with the investigators.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2858-Ib-02
Record Dates: First submitted 2022-03-01; First posted 2022-03-02 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-03

CONDITIONS: Advanced High-grade Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2858 injection (Experimental): TQB2858 injection (1800mg intravenous(iv), on day 1 of every 3 weeks)
  Interventions: Drug: TQB2858 injection

INTERVENTIONS:
Drug: TQB2858 injection — TQB2858 is a dual-function fusion protein that is aProgrammed cell death 1 ligand 1 (PD-L1)/transforming growth factor-β(TGF-β) double antibody.

SUMMARY:
This study is a single-arm, open-label, multicenter Phase Ib clinical trial evaluating TQB2858 injection in the treatment of advanced high-grade sarcoma. To evaluate the preliminary efficacy and safety of TQB2858 injection in patients with advanced high-grade sarcoma, and to explore the relevant biomarkers of TQB2858 injection.

ELIGIBILITY:
Inclusion Criteria:

* 1 Histologically confirmed unresectable, recurrent or metastatic high-grade sarcoma;
* 2 Received at least first-line therapy before, disease progression or intolerance during treatment, or disease progression after treatment; (excluding alveolar soft tissue sarcoma and clear cell sarcoma)

  1. Cohort 1: newly treated acinar soft tissue sarcoma;
  2. Cohort 2: Acinar soft tissue sarcoma with failed PD-1 therapy;
  3. Cohort 3: Other subtypes (pleomorphic sarcoma, classic osteosarcoma, Ewing sarcoma, chondrosarcoma, dedifferentiated liposarcoma, etc.).
* 3 Age: 18 to 70 years old;
* 4 The Eastern Cooperative Oncology Group (ECOG) score: 0 to 1;
* 5 The expected survival period is ≥3 months;
* 6 Normal function of major organs
* 7 Women of childbearing age should agree to use effective contraceptive measures during the study period and 6 months after the end of the study, and have a negative serum or urine pregnancy test within 7 days before enrollment in the study; men should agree to use effective contraception during the study period and after the end of the study period 6 Effective contraceptive measures must be used within one month.
* 8 Patients voluntarily enroll in this study, sign an informed consent form and comply well.

Exclusion Criteria:

* 1 Combined diseases and medical history:

  1. Have presented with or currently have concurrent other malignancies within 2 years.
  2. Unresolved toxic reactions due to any prior treatment above Common Terminology Criteria for Adverse Events (CTCAE) grade 1, excluding alopecia, peripheral sensory nerve disorders.
  3. Major surgical treatment or significant traumatic injury within 28 days prior to the start of study treatment.
  4. Long-term untreated wounds or fractures.
  5. An arterial/venous thrombotic event within 6 months, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism.
  6. Persons with a history of psychotropic substance abuse who are unable to abstain or have a mental disorder.
  7. Subjects with any severe and/or uncontrollable disease, including:
* 2 Tumor-related symptoms and treatment:

  1. Received surgery, chemotherapy, radiotherapy, or other anticancer therapy within 4 weeks prior to the start of study treatment;
  2. Treatment with proprietary Chinese medicines with clear antitumor indications in the National Medical Products Administration (NMPA)-approved drug formulary within 2 weeks prior to the start of study treatment.
  3. Uncontrolled pleural effusions, pericardial effusions, or ascites that still require repeated drainage;
  4. Brain metastases with less than 4 weeks of stable symptom control after discontinuation of dehydrating agents and steroids.
* 3 Research and treatment related:

  1. History of live attenuated vaccination within 28 days prior to the start of study treatment.
  2. Prior history of severe allergy to macromolecular drugs or allergy to known components of TQB2858 injection.
  3. Active autoimmune disease requiring systemic therapy that occurred within 2 years prior to the start of study treatment.
  4. Diagnosis of immunodeficiency or being treated with systemic glucocorticoids or any other form of immunosuppressive therapy.
* 4 Participation in other clinical trials of antineoplastic drugs within 4 weeks prior to enrollment.
* 5 Subjects who, in the judgment of the investigator, have a concomitant illness that seriously jeopardizes the safety of the subject or interferes with the completion of the study, or for whom other reasons are deemed to exist for ineligibility for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 48 weeks
  Objective response rate refers to the percentage of complete response (CR) or partial response (PR) subjects determined by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or modified RECIST1.1 for immune based therapeutics (iRECIST) (CR and PR under iRECIST criteria can occur after imaging disease progression).

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 48 weeks
  Disease control rate refers to the percentage of subjects with CR, PR, or stable disease (SD) of 6 weeks or more as determined by RECIST 1.1 or iRECIST (CR, PR, SD under iRECIST criteria can occur after imaging disease progression).
Overall survival (OS) | Baseline up to die
  Overall survival defined as the time from enrollment to death from any cause.
Progression-Free Survival (PFS) | up to 48 weeks
  PFS will be defined as median number of months from the date of randomization until the first documented sign of disease progression or death due to any causes, whichever occurs first.
Duration of Response (DOR) | up to 48 weeks
  DOR will be defined as median number of months from date of first documented objective response until first documented sign of disease progression or death due to any causes.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China